CLINICAL TRIAL: NCT06828861
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study of ARD-101 for the Treatment of Hyperphagia in Patients With Prader-Willi Syndrome
Brief Title: ARD-101 for Treatment of PWS: The Hunger Elimination or Reduction Objective Trial
Acronym: HERO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aardvark Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVK-101-301
Record Dates: First submitted 2025-02-13; First posted 2025-02-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-05

CONDITIONS: Hyperphagia; Prader-Willi Syndrome
Keywords: Prader-Willi Syndrome; ARD-101; PWS; Prader-Willi; Prader Willi; Prader Willi Syndrome
MeSH Terms: conditions — Hyperphagia; Prader-Willi Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A (Experimental): ARD-101
  Interventions: Drug: ARD-101
- Treatment Arm B (Placebo Comparator): Placebo for ARD-101
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 200 mg BID (twice per day) for 1 week, 400 mg BID for 1 week, 800 mg BID for 10 weeks
  Arms: Treatment Arm B
Drug: ARD-101 — 200 mg BID (twice per day) for 1 week, 400 mg BID for 1 week, 800 mg BID for 10 weeks
  Arms: Treatment Arm A

SUMMARY:
The goal of this clinical trial is to learn if ARD-101 works to treat hyperphagia-related behavior in patients with Prader-Willi syndrome (PWS). It will also teach us about the safety of ARD-101.

The main questions it aims to answer are:

* Does ARD-101 improve the total score of the HQCT-9 (hyperphagia questionnaire for clinical trials, 9 questions)?
* What medical problems do participants have when taking ARD-101?

Researchers will compare ARD-101 to a placebo (a look-alike substance that contains no drug) to see if ARD-101 works to treat hyperphagia in PWS subjects.

Eligible participants will:

* Take ARD-101 or a placebo every day for 12 weeks.
* Visit the clinic or have a tele-visit once every 2 to 4 weeks during dosing and then have a tele-visit 4 weeks after stopping the ARD-101 or placebo.
* Patients/Caregivers will keep a daily diary.

Participants who complete the study may be eligible to enter an open-label extension study where everyone will receive ARD-101.

ELIGIBILITY:
Inclusion Criteria:

* Documented confirmation of Prader-Willi Syndrome (PWS)
* Stable care setting with same, single designated caregiver for at least 6 months prior to Visit 1
* At least 7 years of age or older in the US at the time of consent
* At least 10 years of age or older in Australia
* At least 13 years of age or older in countries outside of the US and Australia

Exclusion Criteria:

* Diagnosis of schizophrenia, bipolar disorder, personality disorder or other severe mood, anxiety or eating disorder (other than hyperphagia).
* Presence of any malignancy within 5 years with the exception of basal or squamous cell carcinoma of the skin, in situ carcinoma of the service, or in situations prostate cancer.
* Presence of clinically relevant renal, hepatic, pancreatic, cardiovascular, neurological, psychiatric, hematological, pulmonary, or GI abnormality that, in the opinion of the investigator, may preclude the patient from safe completion of the study
* Adults: systolic blood pressure >=160 mmHg and/or diastolic blood pressure >=100 mmHg
* Children and Adolescents: systolic blood pressure >=140 mmHg and/or diastolic blood pressure >=90 mmHg.
* Type 1 diabetes mellitus; HbA1c >8.5%
* Use of agents to promote weight gain or loss, alter hunger or appetite within 30 days of Visit 1 and throughout the study.
* Use of any commercially available medication for the treatment of hyperphagia (i.e., Vykat) within 60 days of randomization and throughout the study.
* Very high doses of glucocorticoids in the previous 3 months of Visit 1 and throughout the study.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Hyperphagia Questionnaire for Clinical Trials (HQ-CT) Score | Baseline to Week 12
  The HQ-CT score is a 9 question, 5-point scale to describe the PWS patient's hyperphagia food-related problem behaviors. It is completed by the patient's caregiver. Each question is scored from 0 to 4. The minimum total score is 0 (hyperphagia related behavior symptoms not exhibited) and the maximum total score is 36 (hyperphagia related behavior symptoms are observed).

SECONDARY OUTCOMES:
Change in Caregiver Global Impression of Severity (CaGI-S) for Hyperphagia in Prader-Willi patients | Baseline to Week 12
  The CaGI-S is a single-item, 7-point scale to describe the severity of the PWS patient's hyperphagia (excessive hunger). It is completed by the patient's caregiver. The minimum score is 1 (not present) and the maximum score is 7 (extremely severe). A higher score indicates a worse severity of hyperphagia.
Change in Clinical Global Impression of Severity (CGI-S) Score for Hyperphagia in Prader-Willi patients | Baseline to Week 12
  The CGI-S is a single-item, 7-point scale designed to assess the severity of the PWS patient's hyperphagia (excessive hunger). It is assessed by the clinician and considers the clinician's experience with the PWS population. The minimum score is 1 (normal, not at all ill) and the maximum score is 7 (among the most extremely ill patients). A higher score indicates a worse severity of hyperphagia.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (17):
  - Children's of Alabama, Birmingham, Alabama
  - Rady Children's Hospital, Encinitas, California
  - Children's Hospital of Orange Country, Orange, California
  - Stanford Children's Health Specialty Services, Palo Alto, California
  - Children's Hospital Colorado, Denver, Colorado
  - Nemours Children Clinic Wilmington, Wilmington, Delaware
  - UF Shands Children's Hospital, Gainesville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Maimonides Medical Center, Brooklyn, New York
  - NYU Langone Children's Ambulatory Care Center, Mineola, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Valley Clinical Research, LLC, Weslaco, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
- Canada (4):
  - Alberta Children's Hospital Research Institute, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children's Hospital at London Health Sciences Centre, London, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- South Korea (3):
  - Samsung Medical Center, Seoul, South Korea
  - Inha University Hospital, Incheon
  - Ajou University Hospital, Suwon
- United Kingdom (4):
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - Fulborn Hospital, Cambridge
  - Royal Hospital for Children (Glasgow) - PPDS - PIN, Glasgow
  - The Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: No